CLINICAL TRIAL: NCT01935856
Title: A Dose Escalation, Single and Multiple Dose, Phase 1/2 Study of KHK7580 for Secondary Hyperparathyroidism in Patients Receiving Hemodialysis
Brief Title: Phase 1/2 Study of KHK7580 for Secondary Hyperparathyroidism in Patients Receiving Hemodialysis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7580-003
Record Dates: First submitted 2013-09-02; First posted 2013-09-05 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Hyperparathyroidism
Keywords: patients; receiving; hemodialysis; Secondary
MeSH Terms: conditions — Hyperparathyroidism; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KHK7580 (Experimental)
  Interventions: Drug: KHK7580

INTERVENTIONS:
Drug: KHK7580 — Oral administration

SUMMARY:
This study is designed to evaluate safety, pharmacokinetics and pharmacodynamics after single and multiple administration of KHK7580 for secondary hyperparathyroidism in patients receiving hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Stable chronic renal disease patients receiving hemodialysis 3 times weekly for at least 12 weeks prior to the screening
* intact PTH value ≥ 240 pg/mL at the screening
* Corrected serum calcium ≥ 8.4 mg/dL at the screening

Exclusion Criteria:

* Patients with primary hyperparathyroidism
* Patients who received cinacalcet within 2 weeks prior to the screening
* Patients with change in dose or dosing regimen of active vitamin D/ its analogs, phosphate binders and/or calcium containing compounds within 2 weeks prior to the screening
* Patients who received parathyroidectomy and/or parathyroid intervention
* Patients with uncontrolled hypertension and/or diabetes
* Patients with severe heart disorder
* Patients with severe hepatic disease
* Patients who take investigational drug in other clinical trial within 12 weeks prior to the screening
* Patients who have been judged ineligible to participate in the study by the investigator

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The safety of KHK7580 assessed by number and types of adverse events, laboratory tests, vital signs, electrocardiogram and ophthalmic examination | For 19 weeks
  The safety of KHK7580 assessed by number and types of adverse events, laboratory tests, vital signs, electrocardiogram and ophthalmic examination

SECONDARY OUTCOMES:
Profiles of pharmacokinetics | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72 hours post each single dosing, and pre-dose in Day 1, 3, 5, 8, 12 and 15 in multiple dose period
  Pharmacokinetic parameters such as Maximum concentration (Cmax), time to maximum concentration (tmax), area under the curve (AUC), half-life (t1/2), and etc., are assessed.
Profiles of pharmacodynamics | For 4-15 days after every dosing
  intact PTH, whole PTH, corrected serum calcium, phosphorus, intact FGF23, ionized calcium, calcitonin

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Tokyo, Japan